CLINICAL TRIAL: NCT03642054
Title: Advanced Biomarker Assessment of Adipose Derived Stem Cells and Fibroblasts in Patients With and Without Pelvic Organ Prolapse
Brief Title: Advanced Biomarker Assessment in Pelvic Organ Prolapse
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Johnny Yi, Principal Investigator, Mayo Clinic
Other Study IDs: 17-009172
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-08

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Adipose Derived Stem Cells Fibroblast Stem Cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pelvic Organ Prolapse: Patients having vaginal hysterectomy who demonstrate grade III-IV uterovaginal prolapse.
- Non Pelvic Organ Prolapse: Patients having vaginal hysterectomy who do not demonstrate uterovaginal prolapse.

SUMMARY:
This study will assess advanced biomarkers in patients with and without vaginal prolapse. Assessments will be directed at vaginal fibroblasts and adipose derived stem cells.

DETAILED DESCRIPTION:
Vaginal biopsies and abdominal adipose harvest will be accomplished in patients undergoing vaginal hysterectomy for non-prolapse benign conditions (6) and pelvic organ prolapse (6). Samples of tissues will be divided and portions will be snap-frozen, placed into transport medium for subsequent tissue digestion, and receive paraffin processing. Cells in transport medium will be transported to the Mayo Collaborative Research building (lab of Dr. David Lott) for isolation of fibroblasts and adipose derived stem cells.

The other samples will be transported to the lab of Dr. Andre van Wijnen (RST) to isolate RNA and protein for mRNA, microRNA and additional protein analysis.

Isolated fibroblasts and ASC's from the lab of Dr. Lott (MCA) will be expanded and passaged 3-5 times. ASCs phenotype will be confirmed by flow cytometry. Cells lines will be duplicated and biobanked at the Mayo Clinic Rochester Biotrust and separately biobanked at the Arizona State University lab of scaffold collaborator, Dr. Stephen Massia. Additional frozen cell lines will transported to the lab of Dr. Andre van Wijnen for further processing. . All cells and materials will be used for testing and to advance the science of regenerative medicine. No biobanked cells or materials from this specific project will be used for any future intervention or treatment in humans.

ELIGIBILITY:
Inclusion Criteria-

* Patients undergoing vaginal hysterectomy for non-prolapse benign conditions and pelvic organ prolapse
* at least 18 years old
* Mayo Clinic patient

Exclusion Criteria-

°Patients who have a history of a recognized classic connective tissue disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Undergoing a vaginal hysterectomy for either a pelvic organ prolapse or a non-prolapse benign condition.
Study Population: 6 patients with pelvic organ prolapse and 6 patients without pelvic organ prolapse.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2020-05-18 (Actual)

PRIMARY OUTCOMES:
Advanced biomarker assessments will include messenger RNA sequencing. | one year
  RNA-Seq will determine if there are differences in mRNA or exon expression between cells from prolapse and normal patients, with focus on genes involved in connective tissue metabolism (e.g., collagens, MMPs, TIMPs, myofibroblast markers).

SECONDARY OUTCOMES:
2. Assess 3-D Biomaterial nanoscaffolds as potential carriers of ASC's to treat prolapse. | 1.5 years
  mRNA levels of ASC's in normal and prolapse patients will be assessed as markers for successful cell seeding on 3D-biomaterial nanoscaffolds and compared to cells under standard 2D-cell culture conditions that are used to generate clinical grade ASC's.

CONTACTS AND LOCATIONS:
Overall Officials: Johnny Yi, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Phoenix, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials